CLINICAL TRIAL: NCT03532334
Title: Comparison of 133Xe Scintigraphy With 19F MRI for Evaluation of Lung Ventilation Function: A Non-Inferiority Comparison (DIAL1001007)
Brief Title: Comparison of 133Xe Scintigraphy With 19F MRI
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: unable to accrue in subjects in a timely fashion
Sponsor: Hal C Charles (Other)
Responsible Party: Sponsor-Investigator, Hal C Charles, Assistant Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00089045
Record Dates: First submitted 2018-04-18; First posted 2018-05-22 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Lung Diseases
Keywords: 19F MRI gas Ventilation; 133 XE ventilation Scintigraphy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Perfluorinated Gas/Oxygen Mixture — 19-Fluorine (19F) MRI of the lungs with 21%/79% Oxygen/Perfluorinated Gas, ≤ 25 liters, gas, single visit, < 1 hour
  Other Names: Perfluorinated Propane Imaging

SUMMARY:
The central hypothesis and current observation is that PFx gases used as contrast agents readily provide functional images of the lung airways including important regional ventilation information such as ventilation defect severity and gas trapping. This is a pilot proof of concept study to demonstrate the non-inferiority of 19F MRI gas Ventilation imaging compared to 133Xe ventilation Scintigraphy in subjects with lung disease. The secondary goal of the study is to develop sufficient information to adequately power a pivotal trial of 19F MRI gas Ventilation imaging compared to 133Xe Ventilation Scintigraphy

DETAILED DESCRIPTION:
Aim 1: Compare measures of lung ventilation performance obtained using 133Xe Scintigraphy with performance using 19F Perfluorinated gas MRI using two independent readers.

133Xe Scintigraphy will be scored using the methods described in the statistics section and 19F images will be scored using the methods described in the statistics section. Scores for each subject will be earluated for consistency between readers and modalities. 60% concordance will be considered equivalent.

The outcomes of the work proposed is expected to show the non-inferiority of 19F Perfluorinated gas MRI to 133Xenon Scintigraphy

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial

1. Outpatients of either gender, age > 18.
2. Willing and able to give informed consent and adhere to visit/protocol schedules. (Consent must be given before any study procedures are performed.)
3. Women of childbearing potential must have a negative urine pregnancy test. This will be confirmed before participation in this investigational protocol.
4. Completion of 133Xe ventilation scintigraphy after referral for ventilation imaging for any reason in Pro00081987 A Comparison of Technegas® and Xenon 133 Planar Lung Imaging in Subjects Referred for Ventilation Scintigraphy. The MRI will be accomplished in a timely fashion after the Scintigraphy study based on scheduling availability in the Center for Advanced Magnetic Resonance Development (CAMRD).

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 19F MRI compared to 133 Xenon Scintigraphy | 24 months
  To evaluate the non-inferiority of 19F Perfluorinated gas MRI compared to 133 Xenon Scintigraphy ventilation imaging studies two readers will be selected as having experience reading Xe-133 ventilation scans. Readers will also receive training on interpretation of 19F ventilation images We note that the nature of the images both nuclear medicine and 19F MRI preclude blinding of the readers to the image modality. Images from each modality will be assessed independently and the images will be coded so that readers will not know which image set is from each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Charles, PhD, Principal Investigator — Duke University Medical Center, Department of Radiology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States